CLINICAL TRIAL: NCT02477280
Title: Effects of Expectation, Medication and Placebo on Objective and Self-rated Performance During the Quantified Behavior Test in Patients With Untreated ADHD and Substance Use Disorder
Brief Title: Effects of Expectation, Medication and Placebo on Objective and Self-rated Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Lennart Jansson, PhD RegPsychologist, Region Västmanland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015-03-10/11; 2014-001488-11 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-22 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Substance Use Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): Methylphenidate 20 mg Tablet single-dose per os
  Interventions: Drug: Methylphenidate; Drug: Placebo
- Placebo (Placebo Comparator): Placebo 20 mg Tablet single-dose per os
  Interventions: Drug: Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Cross-over
  Other Names: Medikinet
Drug: Placebo — Medikinet
  Other Names: Medikinet

SUMMARY:
Aim: The purpose of the study is to examine the effects of medication, placebo and expectation on objective and self-rated performance of ADHD core signs during the Quantified Behavior Test in patients with untreated ADHD and substance Use Disorders.

Subjects: Participants are 40 consecutive patients remitted to a neuropsychiatric investigation at the Dependence Clinic Västmanland, Västerås, Sweden.

Method: The study is a double-blind, randomized, placebo-controlled, cross-over study. The study is taken place during four hours on two investigating days, separated by a 4 days wash-out period.

All patients participate on two occasions: In one session they receive the Methylphenidate (MPH) condition, and in the other session they receive the placebo condition. MPH and placebo conditions are counterbalanced across subjects such that half of the participants receive MPH first, and half receive placebo first. Neither the patient nor the research assistant is aware when the participant receive the MPH condition or the placebo condition.

On each investigating day the participant accomplish Questionnaires (Visual Analogical Scales) concerning; (a) expectation, (b) self-rated performance, (c) exhausting exercise, (d) perceived help from the pill and (e) self-rated symptoms. In addition the participant completed A Quick Test of Cognitive Speed (AQT) and two separate Quantified Behavior Test Plus (QbTest) without medication vs MPH/Placebo. QbTest aims to provide objective information regarding core-symptoms of ADHD; hyperactivity on the basis of motor-activity measured with the camera, and inattention and impulsivity on basis of the CPT-test.

DETAILED DESCRIPTION:
Introduction: During the last decade, neuropsychiatric impairments in adults have more often been observed. Requests for neuropsychiatric investigations, especially concerning Attention Deficit Hyperactivity Disorder (ADHD) has increased. The core ADHD symptoms in adults include a frequent and persistent pattern of inattention/distractibility and/or hyperactivity/impulsivity (Adler 2004; Adler & Chua 2002; McGough & Barkley 2004). In a Swedish study, 22 % of the outpatients in general psychiatric care, were diagnosed with ADHD (Nylander et al 2009).

Individuals with ADHD also have an increased risk for other psychiatric disorders, e.g. major depressive episodes, bipolar disorder, anxiety disorders and antisocial personality disorder (Rasmussen & Levander 2009; Torgersen, Gjervan & Rasmussen 2006). The co-occurrence of ADHD and substance use disorder (SUD) is a prevalent phenomenon that has been demonstrated in numerous studies over the past decade (Arias et al 2008; Bernardi et al 2012; van Emmerik-van Oortmerssen et al 2012).

The prevalence of substance abuse in adults with ADHD has been estimated at 50 % and among addicts seeking treatment, one third of the patients are identified as probable ADHD, when screening instruments have been used (Sullivan & Rodnik-Levin 2001; Ohlmeier et al 2008). The National Board of Health and Welfare in Sweden noted that the presence of people with ADHD and substance abuse varies between 20 % and 35 % depending on what kind of drugs that have been used (Socialstyrelsen 2002).

Pharmacotherapy, mainly with central stimulant medication, is considered to be the treatment of choice for ADHD. In addition, there are patients who request an ADHD diagnosis to obtain drug treatment (Harrison, Edwards & Parker 2007).

Patients' expectation can influence the outcome of a treatment (Bingel et al 2011). Linde et al showed that patients with high expectations before the acupuncture treatment, achieved better treating result than the patients who had lower expectations of treatment (Linde, Fässler & Meissner 2011). A person's expectation is an important part of the so-called placebo effect . The placebo effect is well known and clinically important phenomenon in the patient's treatment. Extensive research has been conducted to elucidate this (Meissner et al 2011; Collocca et al 2013; Enck et al 2013).

Patients with substance syndrome often have other expectations for the drug compared to patients with other diagnoses. Some of these patients have often learned to deal with awkward and difficult life situations using drugs (Whalen & Henker 1976; Pelham & Lang 1993). This may increases the risk that the person receives a low confidence in their own ability to solve critical situations without drugs. Therefore, it is important to identify those patients in order to give them a treatment specialized to their need.

This study intends to investigate whether the patient's expectation of their own ability to solve problems increases when they take a drug.

Aim: The purpose of the study is to examine the effects of medication, placebo and expectation on objective and self-rated performance of ADHD core signs during the Quantified Behavior Test in patients with untreated ADHD and substance Use Disorders.

This leads to the following questions ;

1. Does the participant's self-rated expectation of future performance change in the presence of active drug or placebo?
2. Does the participant's self-rated performance change in the presence of active drug or placebo?
3. Does the participant's perception of exertion change in the presence of active drug or placebo?
4. Does the participant's performance on the core signs, Hyperactivity, Inattention and Impulsivity on the QbTest change in the presence of active drug or placebo ?
5. Does the participant's experience of the tablet's efficacy change in the presence of active drug or placebo?

Method: The study is a double-blind, randomized, placebo-controlled, cross-over study. The study is taken place during four hours on two investigating days, separated by a 4 days wash-out period.

Subjects: Participants are 40 consecutive patients remitted to a neuropsychiatric investigation at the Dependence Clinic Västmanland, Västerås, Sweden.

Instruments The Quantized Behavior Test (QbTest) can be included as part of an neuropsychiatric investigation. QbTest measures the three core signs of ADHD, hyperactivity, inattention and impulsivity.

The QbTest combines a Continuous Performance Test (CPT) installed as a software program on a computer with measures of attention and impulsivity and an activity test with measures of motor-activity during 20 minutes. While performing the CPT-test on the computer, movements of the participant are recorded using an infrared camera following a reflective marker attached to a head-band. The CPT-test involves rapid presentations of figures with various shapes (square or circle) and colors (red or blue) and the participant are instructed to press a handheld button when a stimuli subsequently repeats itself (a target) and not to press the button when the stimulus varies relative to the previous one (a non-target). The stimuli are presented at a pace of one per two seconds, each one visible for 200 milliseconds, and the total number of stimuli is 600, presented with a 25% target probability (Knagenhjelm & Ulberstad 2010).

The clinical documentation for QbTest is extensive. Lis et al demonstrated that patients with ADHD were significantly different in the variables of attention and activity from a control group of healthy individuals (Lis et al 2010). Edebol showed that QbTest has a sensitivity of 83 % and a specificity of 57% to detect ADHD in adults (Edebol et al 2011).

The discriminative validity was tested and the results show that QbTest differ not only between those with ADHD and healthy controls , but between clients with ADHD and other clinical groups (Söderström, Pettersson & Nilsson 2014; Edebol, Helldin & Norlander 2012). QbTest has also shown good results as an objective method for monitoring drug treatment with methylphenidate (Ginsberg, Hirvikoski & Grann 2012; Edebol, Helldin & Norlander 2013; Bijlenga & Henker 2014).

The Quick Test measure processing speed and automaticity of naming shapes and colours, Cognitive shifts between visual dimensions and semantic fields and Activation of working memory for processing and monitoring. AQT's objective measures are based on clocked total-naming time. Highly reliable (r = .88 - 96) over time and consistent over repeated trials.

Procedure:

All patients participate on two occasions: In one session they receive the Methylphenidate (MPH) condition, and in the other session they receive the placebo condition. MPH and placebo conditions are counterbalanced across subjects such that half of the participants receive MPH first, and the other half of the participants receive placebo first. Neither the participant nor the research assistant is aware when the participant receive the MPH condition or the placebo condition.

On each investigating day the participant accomplish Questionnaires (Visual Analogical Scales) concerning; (a) expectation, (b) self-rated performance, (c) exhausting exercise, (d) perceived help from the pill and (e) self-rated symptoms. In addition the participant completed A Quick Test of Cognitive Speed (AQT) and two separate Quantified Behavior Test Plus (QbTest) without medication vs MPH/Placebo.

Analyses In this study, hyperactivity has been operationalized with the parameter called "distance", i.e., the length of the path in metres describing the movement of the headband reflector during the test period. Inattention is operationalized on the basis of omission errors. An omission error occurs when no response is registered when the stimulus was a Target, i.e. the button was not pressed when it should have been. Impulsivity is operationalized on the bases of commission errors. A commission error occurs when a response is registered when the stimulus was a Non-Target, i.e. the handheld button is pressed when it should not have been pressed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older.
* ADHD is diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5 criteria).
* Substance Use Disorder is diagnosed according to DSM-5 criteria.
* Qb-score 1.3 or higher on at least one of the weighted summary parameters QbActivity, QbInattention or QbImpulsivity on the QbTest.
* Participants are given their written informed consent to participate in the study.

Exclusion Criteria:

* Affected by alcohol or drugs during the last month.
* Untreated severe comorbid psychiatric or somatic illness.
* Bloodpressure 150/95 or higher.
* Irregular pulse, or pulse 100 or higher.
* No counter indications according to the Medikinet pill.
* Concurrent clinical diagnosis that significantly could affect test performance.
* Concurrent prescription of medicines for ADHD or medicines that significantly could affect test performance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-09; Primary Completion 2021-06 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Change in Weighted summary parameter QbInattention score on the QbTest. | Baseline, 2 hours
  Evaluating change in weighted summary parameter QbInattention score on the QbTest.

SECONDARY OUTCOMES:
Change in Weighted summary parameter QbActivity score on the QbTest. | Baseline, 2 hours
  Evaluating change in weighted summary parameter QbActivity score on the QbTest.
Change in Weighted summary parameter QbImpulsivity score on the QbTest. | Baseline, 2 hours
  Evaluating change in weighted summary parameter QbImpulsivity score on the QbTest.
Change in Self-rated expected performance on the QbTest assessed by a Visual Analogue Scale. | Baseline, 2 hours
  Evaluating change in self-rated expected performance on the QbTest.
Change in Self-rated mental effort during the QbTest assessed by a Visual Analogue Scale. | Baseline, 2 hours
  Evaluating change in self-rated mental effort during the QbTest.
Change in Self-rated severety of the task on the QbTest assessed by a Visual Analogue Scale. | Baseline, 2 hours
  Evaluating change in self-rated severity of the task on the QTest.
Change in Self-rated experienced performance on the QbTest assessed by a Visual Analogue Scale. | Baseline, 2 hours
  Evaluating change in self-rated performance on the QbTest.
Change in Self-rated help from the pill during the QbTest assessed by a Visual Analogue Scale. | Baseline, 2 hours
  Evaluating change in self-rated help from the pill during the QbTest.

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Jansson, PhD, Principal Investigator — Region Västmanland
Locations (1):
- Landstinget Västmanland, Västerås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler LA. Clinical presentations of adult patients with ADHD. J Clin Psychiatry. 2004;65 Suppl 3:8-11. PMID 15046529
- [Background] Adler LA, Chua HC. Management of ADHD in adults. J Clin Psychiatry. 2002;63 Suppl 12:29-35. PMID 12562059
- [Background] Arias AJ, Gelernter J, Chan G, Weiss RD, Brady KT, Farrer L, Kranzler HR. Correlates of co-occurring ADHD in drug-dependent subjects: prevalence and features of substance dependence and psychiatric disorders. Addict Behav. 2008 Sep;33(9):1199-207. doi: 10.1016/j.addbeh.2008.05.003. Epub 2008 May 13. PMID 18558465
- [Background] Bernardi S, Faraone SV, Cortese S, Kerridge BT, Pallanti S, Wang S, Blanco C. The lifetime impact of attention deficit hyperactivity disorder: results from the National Epidemiologic Survey on Alcohol and Related Conditions (NESARC). Psychol Med. 2012 Apr;42(4):875-87. doi: 10.1017/S003329171100153X. Epub 2011 Aug 16. PMID 21846424
- [Background] Bijlenga D, Jasperse M, Gehlhaar SK, Sandra Kooij JJ. Objective QbTest and subjective evaluation of stimulant treatment in adult attention deficit-hyperactivity disorder. Eur Psychiatry. 2015 Jan;30(1):179-85. doi: 10.1016/j.eurpsy.2014.06.003. Epub 2014 Aug 27. PMID 25172155
- [Background] Bingel U, Wanigasekera V, Wiech K, Ni Mhuircheartaigh R, Lee MC, Ploner M, Tracey I. The effect of treatment expectation on drug efficacy: imaging the analgesic benefit of the opioid remifentanil. Sci Transl Med. 2011 Feb 16;3(70):70ra14. doi: 10.1126/scitranslmed.3001244. PMID 21325618
- [Background] Colloca L, Klinger R, Flor H, Bingel U. Placebo analgesia: psychological and neurobiological mechanisms. Pain. 2013 Apr;154(4):511-514. doi: 10.1016/j.pain.2013.02.002. Epub 2013 Feb 13. No abstract available. PMID 23473783
- [Background] Edebol H; Helldin L; Holmberg E; Gustafsson S-A; Norlander T. In search for objective measures of hyperactivity, impulsivity and inattention in adult attention deficit hyperactivity disorder using the Quantified Behavior Test Plus. Europe´s Journal of Psychology 2011, 7, 443-457.
- [Background] Edebol H, Helldin L, Norlander T. Objective Measures of Behavior Manifestations in Adult ADHD and Differentiation from Participants with Bipolar II Disorder, Borderline Personality Disorder, Participants with Disconfirmed ADHD as Well as Normative Participants. Clin Pract Epidemiol Ment Health. 2012;8:134-43. doi: 10.2174/1745017901208010134. Epub 2012 Nov 2. PMID 23166565
- [Background] Edebol H, Helldin L, Norlander T. The weighed core symptom scale and prediction of ADHD in adults - objective measures of remission and response to treatment with methylphenidate. Clin Pract Epidemiol Ment Health. 2013 Oct 18;9:171-9. doi: 10.2174/1745017901309010171. eCollection 2013. PMID 24265648
- [Background] Enck P, Bingel U, Schedlowski M, Rief W. The placebo response in medicine: minimize, maximize or personalize? Nat Rev Drug Discov. 2013 Mar;12(3):191-204. doi: 10.1038/nrd3923. PMID 23449306
- [Background] Ginsberg Y, Hirvikoski T, Grann M, Lindefors N. Long-term functional outcome in adult prison inmates with ADHD receiving OROS-methylphenidate. Eur Arch Psychiatry Clin Neurosci. 2012 Dec;262(8):705-24. doi: 10.1007/s00406-012-0317-8. Epub 2012 Apr 21. PMID 22526730
- [Background] Harrison AG, Edwards MJ, Parker KC. Identifying students faking ADHD: Preliminary findings and strategies for detection. Arch Clin Neuropsychol. 2007 Jun;22(5):577-88. doi: 10.1016/j.acn.2007.03.008. Epub 2007 May 15. PMID 17507198
- [Background] Linde K, Fassler M, Meissner K. Placebo interventions, placebo effects and clinical practice. Philos Trans R Soc Lond B Biol Sci. 2011 Jun 27;366(1572):1905-12. doi: 10.1098/rstb.2010.0383. PMID 21576148
- [Background] Lis S, Baer N, Stein-en-Nosse C, Gallhofer B, Sammer G, Kirsch P. Objective measurement of motor activity during cognitive performance in adults with attention-deficit/hyperactivity disorder. Acta Psychiatr Scand. 2010 Oct;122(4):285-94. doi: 10.1111/j.1600-0447.2010.01549.x. Epub 2010 Feb 25. PMID 20199487
- [Background] McGough JJ, Barkley RA. Diagnostic controversies in adult attention deficit hyperactivity disorder. Am J Psychiatry. 2004 Nov;161(11):1948-56. doi: 10.1176/appi.ajp.161.11.1948. PMID 15514392
- [Background] Meissner K, Bingel U, Colloca L, Wager TD, Watson A, Flaten MA. The placebo effect: advances from different methodological approaches. J Neurosci. 2011 Nov 9;31(45):16117-24. doi: 10.1523/JNEUROSCI.4099-11.2011. PMID 22072664
- [Background] Nylander L, Holmqvist M, Gustafson L, Gillberg C. ADHD in adult psychiatry. Minimum rates and clinical presentation in general psychiatry outpatients. Nord J Psychiatry. 2009;63(1):64-71. doi: 10.1080/08039480802416323. PMID 18991159
- [Background] Ohlmeier MD, Peters K, Te Wildt BT, Zedler M, Ziegenbein M, Wiese B, Emrich HM, Schneider U. Comorbidity of alcohol and substance dependence with attention-deficit/hyperactivity disorder (ADHD). Alcohol Alcohol. 2008 May-Jun;43(3):300-4. doi: 10.1093/alcalc/agn014. Epub 2008 Mar 7. PMID 18326548
- [Background] Pelham WE; Lang AR. Parental alcohol consumption and deviant child beha-vior: Laboratory studies of reciprocal effects. Clinical Psychology Review 1993, 13, 763-784.
- [Background] Rasmussen K, Levander S. Untreated ADHD in adults: are there sex differences in symptoms, comorbidity, and impairment? J Atten Disord. 2009 Jan;12(4):353-60. doi: 10.1177/1087054708314621. Epub 2008 Mar 26. PMID 18367759
- [Background] Sullivan MA, Rudnik-Levin F. Attention deficit/hyperactivity disorder and substance abuse. Diagnostic and therapeutic considerations. Ann N Y Acad Sci. 2001 Jun;931:251-70. doi: 10.1111/j.1749-6632.2001.tb05783.x. PMID 11462745
- [Background] Soderstrom S, Pettersson R, Nilsson KW. Quantitative and subjective behavioural aspects in the assessment of attention-deficit hyperactivity disorder (ADHD) in adults. Nord J Psychiatry. 2014 Jan;68(1):30-7. doi: 10.3109/08039488.2012.762940. Epub 2013 Mar 26. PMID 23527787
- [Background] Torgersen T, Gjervan B, Rasmussen K. ADHD in adults: a study of clinical characteristics, impairment and comorbidity. Nord J Psychiatry. 2006;60(1):38-43. doi: 10.1080/08039480500520665. PMID 16500798
- [Background] van Emmerik-van Oortmerssen K, van de Glind G, van den Brink W, Smit F, Crunelle CL, Swets M, Schoevers RA. Prevalence of attention-deficit hyperactivity disorder in substance use disorder patients: a meta-analysis and meta-regression analysis. Drug Alcohol Depend. 2012 Apr 1;122(1-2):11-9. doi: 10.1016/j.drugalcdep.2011.12.007. Epub 2011 Dec 30. PMID 22209385
- [Background] Whalen CK, Henker B. Psychostimulants and children: a review and analysis. Psychol Bull. 1976 Nov;83(6):1113-30. No abstract available. PMID 792938